CLINICAL TRIAL: NCT05010447
Title: Feasibility of an Avatar-Led and ACT-Based Smartphone Application for Adjunctive Psychotherapy in In- and Outpatients: Virtual Coach App
Brief Title: Feasibility of an Avatar-Led and ACT-Based App for Adjunctive Psychotherapy in In- and Outpatients: Virtual Coach App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Basel (Other)
Collaborators: Universitäre Psychiatrische Kliniken (UPK) Basel (Unknown); Klinik Sonnenhalde AG Psychiatrie und Psychotherapie (Unknown); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andrew Gloster, Prof. Dr., Division of Clinical Psychology & Intervention Science, University of Basel, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VC
Record Dates: First submitted 2021-07-07; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Mental Disorder
Keywords: Avatar-guided smartphone application; Acceptance and Commitment Therapy; Mental disorders; Device feasibility; Application feasibility
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Micro-Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Participants receive the Virtual Coach App for one week at the beginning of their therapy and one week towards the end of their therapy.
  Interventions: Device: Virtual Coach App

INTERVENTIONS:
Device: Virtual Coach App — The avatar-guided app aims to deepen the user's understanding of Acceptance and Commitment Therapy (ACT) and promote application of ACT skills in every-day-life. Event-Sampling-Methodology (ESM) is used to capture the user's progress as it unfolds.

SUMMARY:
The aim of this study is to test the feasibility of an application for smartphones based on Acceptance and Commitment Therapy (ACT) that was designed to increase treatment adaptation (i.e. learning therapy skills) and treatment utility (i.e. feedback for the patient). The use of this avatar- led application will be tested by patients with mental disorders adjunctive to their therapy. Patients will be given a smartphone for one week with the application developed specifically for this purpose. The study will be a single group design and patients will be assessed two times: before and after having tested the application. Measurements will include acceptability (adherence, utilization, utility, satisfaction) of the application, as well as patients characteristics, such as diagnostic interviews, questionnaires about symptomatology, well-being, social interactions, and an exit questionnaire when leaving the study to assess what was learned.

DETAILED DESCRIPTION:
This study will use a digital tool with the aim to test whether a "Virtual Coach" can increase treatment adaptation (i.e., learning of therapy skills, prevent drop-out), treatment utility (i.e., via direct feedback to the patient and therapist), and increase adherence. The digital tool will be an avatar-led application for smartphones and be based on the Acceptance and Commitment Therapy.

The "Virtual Coach" will be used adjunctive to therapy and help patients initiate behavioral changes and accelerate the learning of new therapy skills. The questions addressed will be the following: a) adherence to and utilization of the Virtual Coach itself ; b) application of therapy skills; c) perceived usefulness of the Virtual Coach by patients and therapists, and d) the frequency of prosocial behaviors and their impact on well-being.

The main purpose of this study is the feasibility of using the Virtual Coach adjunctively to a therapy. However, it also will be explored how outcomes may be related to the severity of symptoms and other factors.

The study contains a pilot test in a single-arm trial to evaluate the main outcomes of acceptability (adherence, utilization, utility, satisfaction) with n = 40. Patients will be assessed at baseline and again after the course of their psychotherapy (post-assessment).

Patients will complete informed consent, undergo a short diagnostic assessment, then receive a smartphone with the application to carry for one week. They will be asked to use the application at least three times per day in order to practice skills involved in the treatment. The assessment targets will include intentions, activities, and goals of the patient, interpersonal activities, and health behaviors. Subjective reports (e.g., emotions, thoughts, reactions, plans) and objective data (response times, adherence to prompts, etc.) will be tracked. In addition to the main acceptability outcomes, additional assessments will be used to measure patient characteristics. This will include a diagnostic interview, questionnaires about symptomatology, well-being, social interactions, and an exit questionnaire when leaving the study to assess what was learned.

ELIGIBILITY:
Inclusion Criteria:

* Current undergoing inpatient or outpatient psychotherapy;
* ability to speak German or English;
* giving informed consent.

Exclusion Criteria:

* not able to take part as assessed by the clinic's medical/therapeutic staff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
User Experience Questionnaire | once at Baseline (beginning of therapy/week 1)
  User Experience Questionnaire (UEQ; Laugwitz, B., Schrepp, M. & Held, T., 2008). The UEQ is a short questionnaire using semantic differentials (word pairs with opposite meanings) to allow for fast and intuitive responses. An example item would be "attractive - unattractive". Items are scored on a 7-point Likert scale and range from full agreement with the negative term (-3) to the full agreement with the positive term (+3). Half of the items start with the positive term, the rest with the negative term. Higher sum scores indicate more positive evaluation of the app.
System Usability Scale | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  System Usability Scale (SUS; adapted from Brooke, 1996) embedded. SUS scores have a range of 0 to 100. A high score indicates a high system usability; and where 1 = strongly disagree and 5 = strongly agree.
Semi-structured User Experience Questionnaire | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  Self-designed questionnaire with closed and open questions regarding the user's experience with the app. Questions were tested in a pilot and then adapted in a feedback round. They include items such as "How was your week with Virtual Coach?", "What about Virtual Coach did you like best?", "What about Virtual Coach did you like least?", etc. The Interview also includes space for open comments from the user.
User Adherence Meta-Variables | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  Metavariables and app-usage of participants are collected automatically while the app is being used by the study participant, such as:
  * Number of prompts responded (where a higher number equals more adherence)
  * Number of prompts finished (where a higher number equals more adherence)
  * Number of exercises completed (where a higher number equals more adherence)
  * Number of additional exercises completed (where a higher number equals more adherence)
  * Time to complete prompts (where the average time of the sample should represent an adequate time for an adherent user to complete the prompt)
  * An answers typed in by the participant in the app during its usage

SECONDARY OUTCOMES:
Therapy Expectancy | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Credibility and Expectancy Questionnaire" (CEQ; adapted from Devilly & Borkovec, 2000). The questionnaire contains 6 items. The first three items for the credibility factor. These items are rated on 9- point scales ranging from 1 (Not at all logical/useful/confident) to 9 (Very logical/useful/confident), with a total score possible range of 3 to 27. The last three items form the expectancy factor: one item is assessed on the same 9-point scale as the credibility items and two are assessed on an 11-point scale (from 0% to 100% in 10-point increments), responses are first standardized before summing to render the expectancy total score. A higher score symbolizes a high expectancy of the patient in the the treatment.
Psychological Flexibility | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "PsyFlex" (Gloster et al., in review). The questionnaire contains 6 items, which refer to the last 7 days. A higher score indicates a higher psychological flexibility. The scale is a 5-point scale, where 5 = very often, 4 = often, 3 = from time to time, 2 = seldom, and 1 = very seldom.
Social Interaction | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Social Interaction Scale" (SIS; self-designed). The Social Interaction Scale is a self-designed 3-item self-report measuring the frequency, duration, and discomfort of social interactions in the last 24 hours. Item one is rated on a 4-point scale, item 2 on a 3-point scale. The SIS has been previously used in a longitudinal study to measure the level of social interaction experienced by the respondent.
Disability | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "World Health Organization Disability Assessment Schedule, WHODAS-2" (Garin et al., 2010).The total score has a range from 0 to 100, with higher scores indicating higher levels of disability. The questionnaire contains 18 items (in the german version) measuring abilities on a 5-point scale where 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, 5 = Extreme or cannot do. In the last three items participant have to indicate the number of days during the last 30 days when they had the difficulties listed in the 15 first items or when participants were unable/restricted to carry out their usual activities or work because of their health condition.
Emotion Dysregulation | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Difficulties in Emotion Regulation Scale" (DERS; Gratz & Roemer, 2004). The measure is scored such that higher scores reflect greater difficulties in emotion regulation. The questionnaire contains overall 36 items and is measured on a 5-point scale, where 1 = almost never (0 - 10%), 2 = sometimes (11 - 35%), 3 = about half the time (36 - 65%), 4 = most of the time (66 - 90%), 5 = almost always (91 -100%). The minimal possible score is 36; the maximum possible score is 180.
Wellbeing | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "The Mental Health Continuum - Short Form" (MHC-SF; Karim & Noor, 2006). The MHC-SF is a 14-item self-report measure of emotional, social and psychological well-being. Each item is rated on a 6-point scale, where never = 0, once or twice = 1, about once a week = 2, about 2 or 3 times a week = 3, almost every day = 4, every day=5. The total score has a thus a range from 0 - 70. A higher score indicates better mental health.
Symptomatology | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Brief Symptom Checklist" (BSCL; Franke et al., 2015). The BSCL represents a psychological test instrument for the assessment of psychological symptoms and psychological distress. The questionnaire contains 53 items, and a 5-point scale is used, where 0 = not at all, 1 = a little, 2 = quite a bit, 3 = a lot and 4 = overwhelmingly. The GSI (Global Severity Index), the PST (Positive Symptom Total), and the PSDI (Positive Symptom Distress Index) are formed as overall scores and can range from 20 to 80. Higher scores indicate higher symptom load.
Perceived Stress | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  The "Daily Stress Scale" (DSS; Scholten et al., 2014) is a 7-item self-report measure of perceived stress in different life domains. The subjective degree of stress is assessed on a 7-point scale from 1 (little incriminating) to 7 (not affected). Higher scores indicate a higher perceived stress level.
Prosocial Behavior | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Prosocialness Scale for Adults" (PSA; Caprara et al., 2005). The Prosocialness Scale for Adults measures an individuals prosocial behavior with 16 items. For all items a five-point Likert scale is used; indicating whether the statement was never/almost never true = 1, occasionally true = 2, sometimes true = 3, often true = 4, and almost always/always true = 5. Higher score indicate a greater markedness of the prosociality trait.
Self-efficacy | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Self-Efficacy Scale" (self-developed). This questionnaire contains two sections with an overall of 7 items. The first four items are measured on a 5-point scale from "not sure at all" (coded as 1) to "very sure" (coded as 5). The last three items are also measured on a 5-point scale with "totally disagree" coded as 1 to "totally agree" coded as 5. Higher scores indicate higher self-efficacy.
Media and Technology Usage and Attitudes | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  "Media and Technology Usage and Attitudes Scale" (MTUAS; Rosen et al., 2013). For all items a five-point Likert scale (strongly agree = 5, agree = 4, neither agree nor disagree = 3, disagree = 2, strongly disagree = 1) was used. Item 15 is the only item, where the scoring was reversed. The first three items as well as item 7,8 and 9 assess positive attitudes towards technology and higher scores indicate more positive attitudes toward technology. The item 4 to 6 measure technological dependency and anxiety. Higher scores indicate a greater technological anxiety and dependence. Item 10 to 12 are part of the scale for negative attitudes with higher scores indicating more negative attitudes toward technology. The last four items (13 to 16) measure a preference for task switching; higher scores indicate a greater preference for task switching.
Trusting Beliefs towards the Avatar | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  Trusting Beliefs is captured by a 10-item rating scale (modified from Wang & Benbasat, 2007) with a 7-point Likert scale, where 1 = totally agree and 7 = totally disagree. Lower scores indicate trusting beliefs towards the Avatar, and higher scores indicate distrust.
Perceived Social Presence of the Avatar | up to 3 months (from Baseline/beginning of treatment to Post/end of treatment)
  Social Presence is captured by a one-item scale (modified from Gefen & Straub, 2003) measuring social presence by a 7-point scale, that is coded as following: 1 = strongly disagree to 7 = strongly disagree. A Lower score a good social presence of the Avatar, a higher score indicates a lack of social presence.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T. Gloster, Prof. Dr., Study Chair — University of Basel, Faculty of Psychology, Division for Clinical Psychology and Intevention Science
Locations (2):
- Switzerland (2):
  - Universitäre Psychiatrische Kliniken (UPK) Basel, Basel, Canton of Basel-City
  - Klinik Sonnenhalde, Riehen, Canton of Basel-City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Kashdan TB, Rottenberg J. Psychological flexibility as a fundamental aspect of health. Clin Psychol Rev. 2010 Nov;30(7):865-78. doi: 10.1016/j.cpr.2010.03.001. Epub 2010 Mar 12. PMID 21151705
- [Background] Karekla M, Savvides SN, Gloster A. An Avatar-Led Intervention Promotes Smoking Cessation in Young Adults: A Pilot Randomized Clinical Trial. Ann Behav Med. 2020 Oct 1;54(10):747-760. doi: 10.1093/abm/kaaa013. PMID 32383736
- [Background] Trull TJ, Ebner-Priemer UW. Using experience sampling methods/ecological momentary assessment (ESM/EMA) in clinical assessment and clinical research: introduction to the special section. Psychol Assess. 2009 Dec;21(4):457-62. doi: 10.1037/a0017653. PMID 19947780